CLINICAL TRIAL: NCT04445194
Title: A Multi-center, Double-blind, Randomized, Placebo Parallel Controlled, Safety and Tolerability Phase I Clinical Trial of Recombinant Novel Coronavirus Vaccine (CHO Cells) in Healthy People Between 18 and 59 Years of Age
Brief Title: Phase I Clinical Study of Recombinant Novel Coronavirus Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCV-Ⅰ-healthy
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Coronavirus
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — Coronavirus Infections | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Population I (Experimental): Population I has 20 subjects and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population I is intramuscular injection of deltoid muscle of upper arm with low dose of vaccine.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell) low-dose group
- Population II (Experimental): Population II has 20 subjects and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population II is a high-dose vaccine intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) high-dose group
- Population Ⅲ (Placebo Comparator): Population Ⅲ has 10 subjects and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population Ⅲ is a placebo intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) low-dose group — Intramuscular injection of deltoid muscle of upper armof 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population I
Biological: Recombinant new coronavirus vaccine (CHO cells) high-dose group — Intramuscular injection of deltoid muscle of upper armof 50μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population II
Biological: Recombinant new coronavirus vaccine (CHO cells) placebo group — Intramuscular injection of deltoid muscle of upper armof 0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population Ⅲ

SUMMARY:
In this trial, a total of 50 subjects were recruited; the test vaccines were divided into 3 groups, low-dose vaccine groups, high-dose vaccine groups, and placebo groups. The first-stage randomized participants in the low-dose group (20 cases) and the placebo group (5 cases) were evaluated for 7 days. After the 7-day safety data was evaluated and agreed by the DSMB, the second-stage study was conducted. Into the high-dose group (20 cases) and placebo group (5 cases) subjects; follow-up to 30 days, after the safety assessment by the investigator and consent, then inoculate the second dose. Observation was performed for 1.0 hour after the second dose. The researchers conducted a safety evaluation and agreed to follow-up after discharge.

DETAILED DESCRIPTION:
In this trial, a total of 50 subjects were recruited; the test vaccines were divided into 3 groups, low-dose vaccine groups, high-dose vaccine groups, and placebo groups. The first-stage randomized participants in the low-dose group (20 cases) and the placebo group (5 cases) were evaluated for 7 days. After the 7-day safety data was evaluated and agreed by the DSMB, the second-stage study was conducted. Into the high-dose group (20 cases) and placebo group (5 cases) subjects; follow-up to 30 days, after the safety assessment by the investigator and consent, then inoculate the second dose. Observation was performed for 1.0 hour after the second dose . The researchers conducted a safety evaluation and agreed to follow-up after discharge.

In this trial, all adverse events (AE), all AEs from 0-7 days, and all AEs from 8-30 days will be collected 30 minutes after each dose, and all AEs will be collected from the first dose to 30 days after the entire vaccination, and the first dose will be inoculated to the full course All serious adverse events (SAE) 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the observation age of this clinical trial: 18-59 years old (both included) adults.
* The subjects themselves voluntarily agreed to participate in the study, and signed an informed consent form, and can provide legal identification; understand and abide by the requirements of the trial protocol; can participate in a half-year follow-up.
* Body temperature under armpit <37.3 ℃.
* Body mass index (BMI) at 18-28kg / m² (inclusive).
* Female and male subjects of childbearing age took effective contraception during the study.

Exclusion Criteria:

* The vital signs, physical examination and laboratory test indicators of the population specified in the plan are abnormal and have clinical significance as determined by the clinician;
* Have a history of severe allergies to any component of the research vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis (Arthus reaction); or any previous History of serious side effects of vaccines or drugs, such as allergies, urticaria, skin eczema, dyspnea, angioedema, etc .
* Those with a history of SARS and COVID-19, meet any of the following:

  1. previous history of SARS-CoV and SARS-CoV-2 infection or morbidity;
  2. during the current SARS-CoV-2 epidemic, there is a diagnosis with the new crown Patient / suspected patient contact history;
  3. positive for SARS-CoV-2 IgM and / or IgG antibodies;
  4. positive for real-time fluorescent RT-PCR nucleic acid.
* Have taken antipyretics or painkillers within 24 hours before the first dose of vaccine.
* Inoculate subunit vaccine and inactivated vaccine within 14 days before the first dose of vaccination, and inoculate live attenuated vaccine within 30 days.
* People with the following diseases:

  1. Acute febrile illness;
  2. Digestive system diseases (eg, diarrhea, abdominal pain, vomiting, etc.) in the past 7 days;
  3. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc .;
  4. Congenital or acquired immunodeficiency or autoimmune disease history or within 6 months of receiving immunomodulator treatment, such as hormones; or monoclonal antibodies; or thymosin; or interferon, etc .; but local medications (such as ointment are allowed , Eye drops, inhalation or nasal spray), local administration should not exceed the dosage recommended in the instructions or have any signs of systemic exposure;
  5. The chest imaging examination is clinically significant if the investigator judges that the abnormality is clinically positive, or any positive of hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus HIV antibody or syphilis specific antibody;
  6. Neurological diseases or neurodevelopmental disorders (eg, migraine, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficit, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis ); History of mental illness or family history;
  7. Functional spleenlessness, and spleenlessness or splenectomy for any reason;
  8. There are serious chronic diseases or conditions that cannot be controlled smoothly in the advanced stage, such as diabetes and thyroid disease;
  9. Severe liver and kidney diseases; respiratory diseases that currently require daily medication (eg, chronic obstructive pulmonary disease [COPD], asthma) or any treatment that exacerbates respiratory diseases (eg, exacerbated asthma) within the last 5 years; suffers History of severe cardiovascular disease (such as congestive heart failure, cardiomyopathy, ischemic heart disease, arrhythmia, conduction block, myocardial infarction, pulmonary heart disease) or myocarditis or pericarditis;
  10. have thrombocytopenia, any coagulopathy, or receive anticoagulant treatment, etc .;
  11. Cancer patients;
  12. Have received blood or blood-related products, including immunoglobulin within 3 months; or plan to use it during the study.
* Lactating women or pregnant women (including blood or urine pregnancy test positive).
* Any research or unregistered product (medicine, vaccine, biological product or device) other than the research product was used within 3 months before the application of the test drug / vaccine, or planned to be used during the study.
* People with halo and halo needles.
* The investigator believes that the presence of any disease or condition in the subject may put the subject at an unacceptable risk; the subject cannot meet the protocol requirements; and interfere with the assessment of vaccine response.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | Up to one year after the last vaccination
  The main observation methods of adverse reactions mainly include laboratory examination, local reactions and systemic reactions at the administration site, vital signs, blood routine, blood biochemistry, and urine routine.

SECONDARY OUTCOMES:
Immunogenic end point | Within 6 months after the last dose of vaccination
  All subjects The levels of IL-2, IL-4, IL-5, IL-6 and IFN-γ levels before each vaccination, day 14 after the first vaccination, day 7 after the second vaccination, and 1 and 6 months after the entire vaccination.
  All subjects before each dose of vaccination, on the 14th day after the first dose, on the 7th day after the second and 1 month and 6 months after the full vaccination That Positive rate of New coronavirus (SARS-CoV-2) neutralizing antibody、S protein binding antibody (IgG) and RBD protein binding antibody (IgG).
  All subjects before each dose of vaccination, on the 14th day after the first dose, on the 7th day after the second and 1 month and 6 months after the full vaccination That Titer level and its multiplier than before exemption of New coronavirus (SARS-CoV-2) neutralizing antibody、S protein binding antibody (IgG) and RBD protein binding antibody (IgG).

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, master, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Yang S, Li Y, Dai L, Wang J, He P, Li C, Fang X, Wang C, Zhao X, Huang E, Wu C, Zhong Z, Wang F, Duan X, Tian S, Wu L, Liu Y, Luo Y, Chen Z, Li F, Li J, Yu X, Ren H, Liu L, Meng S, Yan J, Hu Z, Gao L, Gao GF. Safety and immunogenicity of a recombinant tandem-repeat dimeric RBD-based protein subunit vaccine (ZF2001) against COVID-19 in adults: two randomised, double-blind, placebo-controlled, phase 1 and 2 trials. Lancet Infect Dis. 2021 Aug;21(8):1107-1119. doi: 10.1016/S1473-3099(21)00127-4. Epub 2021 Mar 24. PMID 33773111